CLINICAL TRIAL: NCT05426577
Title: Evaluation of Less Invasive Procedures for Visceral Leishmaniasis Treatment Efficacy Monitoring Test of Cure
Acronym: VL-ToC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Leishmaniasis Research and Treatment Cener University of Gondar, Ethiopia (Unknown); WHO Collaborating Centre for Leishmaniasis, INstituto de Salud Carlos III, Spain (Unknown); University of Amsterdam Medical Center, Netherlands (Unknown); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: VL-ToC-AfriKADIA
Record Dates: First submitted 2022-06-01; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Visceral Leishmaniasis
Keywords: leishmania; leishmaniasis; kala azar
MeSH Terms: conditions — Leishmaniasis, Visceral; Leishmaniasis | interventions — Light

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ELISA, LAMP, Cytokine Release Assay — IgG1 ELISA: ELISA that employs soluble Leishmania lysate or protein antigen.Results are recorded as antibody titres, which are measured by the absorbance values of products generated using enzyme conjugated anti-human antibodies.
  Cytokine release assay (CRA): In this assay whole blood is stimulated for 24 hours with leishmania antigen. Cytokine levels are then assessed in the plasma fraction using flow cytometry with the BD™ Cytometric Bead Array for Human Cytokines or standard ELISA kits for human cytokines commercialized by Sigma-Aldrich (RAB0268-IL-2, RAB0222-IFN-g, RAB0224-IL-10, RAB0476-TNF-a, RAB0119-IP-10).
  LAMP test for VL: We will use the LoopampTM Leishmania Detection Kit, CE-marked and produced Eiken Chemical Co., Japan.

SUMMARY:
Left untreated, visceral leishmaniasis (VL) is fatal. The highest burden of VL worldwide is in eastern Africa where field-adapted diagnostic and test-of-cure tools and treatment are lacking. The current laboratory tool to help assessing cure, treatment failure and relapse is microscopy, based on invasive sampling (e.g. splenic or bone marrow aspirate). Non-invasive, more sensitive tools will enable these assessments with minimum risk and discomfort to patients.

This study aims to evaluate immunological and molecular tests to predict cure and relapse, and to replace with these the current invasive methods.

The study will be conducted at the Leishmaniasis Research and Treatment Centre (LRTC), Gondar University Hospital, Ethiopia It will be a non-intervention study, the tools under evaluation will be considered as index tests; their results will not influence patient management during the duration of the study. Patient management will follow the national guidelines for VL diagnosis and management in Ethiopia.

DETAILED DESCRIPTION:
CONTEXT Visceral leishmaniasis (VL), or kala-azar, is caused by parasitic protozoa of the Leishmania donovani species complex, which are transmitted by the bite of infected female phlebotomine sand flies. VL has a worldwide distribution throughout Asia, eastern Africa, South America and the Mediterranean basin. A proportion of infected individuals present with insidiously evolving symptoms, with splenomegaly, irregular fever, anaemia or pancytopaenia, weight loss and weakness, occurring progressively over a period of weeks or even months. And the disease can be fatal without treatment in up to 90% of cases.

In 1990, the worldwide incidence of VL was estimated at 500,000 cases annually. Since then, it has significantly decreased. A WHO report on the 14 high-burden countries (> 100 cases/year) reported 30,758 new cases of VL in 2014, with under-reporting between 1.2- and 4-fold. This drastic reduction in the last decades is largely attributed to a sharp decline in incidence in Southeast Asia, from approximately 50,000 reported cases in 2006-2007, to 10,311 in 2014. A successful elimination campaign, natural fluctuations in incidence and improvements in local living conditions have contributed to the decrease. Currently, the highest burden of VL worldwide is in eastern Africa, where there is a lack of appropriate diagnostic tools and treatment. Most of the cases are observed in Ethiopia, Kenya, Somalia, Sudan, South Sudan and Uganda. Of the six countries currently representing 91% of the overall VL burden worldwide, four are in eastern Africa - Ethiopia, South Sudan, Sudan and Somalia.

With targets for VL elimination being reached in Southeast Asia, the WHO has recently encouraged partners to improve the tools for better control and eventual elimination of VL in specific foci in eastern Africa. Important challenges for disease control include: inconsistent performance of RDTs in different regions; suboptimal efficacy of treatment with potentially toxic injectable medicines; lack of drug resistance monitoring; insufficient access to early diagnosis and treatment; and lack of a test-of-cure and prediction of relapses. All this has a significant impact on morbidity, mortality, loss of quality of life and economic development. We believe that improving access to diagnostic and treatment monitoring tools for VL is the cornerstone of successful VL control/elimination approaches.

New drugs and drug combinations for VL are being evaluated by DNDi and LEAP partners at several study sites, who showed that in Eastern Africa, sodium stibogluconate (SSG) and paromomycine (PM) in combination offer an advantage compared to the previous SSG monotherapy. Close patient monitoring during treatment and follow-up, provides a unique opportunity for evaluating new tools and markers of cure and relapses, as we propose in this study.

STUDY RATIONALE In VL clinical trials, patients fulfilling pre-defined inclusion criteria are enrolled based on diagnosis by Leishmania positive tissue aspirate (spleen, bone marrow or lymph node) and microscopy, which is also the method used as the parasitological test-of-cure at the end of treatment. Although sensitive (variable depending on the tissue sample), this traditional method bears limitations, warranting new improved non-invasive tools. Spleen aspiration and microscopy also have limitations, including difficulty in harmonizing microscopy results, as tissue aspirates are not homogeneous, reflecting inaccurate assessments of parasite load. In many patients, the spleen shrinks with treatment, making monitoring by splenic aspiration at the end of treatment difficult. In these cases, bone marrow aspirates are often analysed for test-of-cure, which makes quantitative comparisons of parasite loads before and after treatment even more difficult. Finally, splenic aspiration is invasive with risk of severe complications.

Diagnosing VL using a sensitive diagnostic test based on peripheral blood is much more favourable. Nucleic acid amplification tests (NAAT) have proven sensitive for detection of Leishmania parasites in blood and have a potential role in the diagnostic algorithm of primary VL. However, in VL endemic settings, most NAAT are restricted to well-equipped laboratories. Recently, FIND, in collaboration with other partners, developed a robust NAAT, loop-mediated isothermal amplification (LAMP) that can be used at the basic laboratory level (e.g. microscopy laboratory). An additional advantage of LAMP is that by using a fluorimeter or turbidimeter, it could reproducibly semi-quantify parasite load, avoiding parasite grading based on microscopy of tissues obtained invasively. The WHO has recently recommended LAMP for the diagnosis of pulmonary tuberculosis.

A top research priority highlighted by the WHO Expert Committee on the Control of Leishmaniasis is identification of a biomarker of treatment failure and relapses, as opposed to cure after chemotherapy [1]. New tools and biomarkers to monitor the immune response of VL patients during therapy, such as immunoglobulin isotypes or cytokines, and that can be used to predict relapses, are important in eastern Africa, given the high relapse rate and that VL/HIV co-infection is a major determinant of relapses [1,3]. New T-cell-based interferon-γ release assays have shown that IFN-γ in Leishmania-stimulated whole blood increases gradually and significantly after successful treatment of patients infected with L. donovani or L. infantum . Whole blood stimulation and cytokine release assay (CRA) and cell proliferation assay (CPA) have demonstrated their usefulness to predict relapses in immunodepressed patients. CRA and IFN-γ analysis helped to confirm cure and risk of relapses in solid organ transplant individuals, while CPA was a good predictive marker of non-appearance of relapses in HIV patients co-infected with Leishmania. On the other hand, with the use of simple serological tests (ELISA), a strong evidence has been presented for the use of anti-Leishmania IgG1 in monitoring treatment outcomes in VL [10]. We propose a collaboration between European and Ethiopian research institutions, with sound expertise on VL, which will capitalize on LEAP's working infrastructure to evaluate the usefulness of an ELISA test detecting anti-Leishmania IgG1 antibodies, Leishmania-specific lymphocyte proliferation, cytokine release assays and LAMP to predict treatment failure and relapse in VL patients.

With targets for VL elimination being reached in Southeast Asia, the WHO has recently encouraged partners to improve the tools for better control and eventual elimination of VL in specific foci in eastern Africa. Important challenges for disease control include: inconsistent performance of RDTs in different regions; suboptimal efficacy of treatment with potentially toxic injectable medicines; lack of drug resistance monitoring; insufficient access to early diagnosis and treatment; and lack of a test-of-cure and prediction of relapses. All this has a significant impact on morbidity, mortality, loss of quality of life and economic development. Improving access to diagnosis and treatment monitoring tools for VL is the cornerstone of successful VL control/elimination approaches.

OBJECTIVES The objective of the proposed study is to evaluate immunological (whole blood cytokine release assay, cell proliferation assay, IgG1 anti-Leishmania) and molecular (loop-mediated isothermal amplification) tests to predict cure and relapse, and to replace with these the current invasive methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical signs and symptoms of VL and confirmatory parasitological microscopic diagnosis.
* Patients for whom written informed consent has been obtained (if aged 18 years and over) or signed by parents(s) or legal guardian for patients under 18 years of age (in the case of minors, assent from the children also needs to be obtained as per country regulatory requirements).

Exclusion Criteria:

VL cases will not be enrolled in the study if any of the following exclusion criteria apply:

* Patients who are cases of VL relapse, post- or para-kala-azar dermal leishmaniasis or who have received any anti-leishmanial drugs within the last six months.
* Patients not eligible for treatment with SSG+PM:

  * Patients with severe malnutrition.
  * Patients with positive HIV diagnosis.
  * Patients with previous history of hypersensitivity reaction or known drug class allergy to any of the study treatments (SSG or PM).
  * Patients with previous history of cardiac arrhythmia or with a clinically significant abnormal ECG.
  * Patients suffering from a concomitant severe infection such as TB or any other serious underlying disease (cardiac, renal, hepatic), or chronic condition which would preclude evaluation of the patient's response to study medication.
* Patients who cannot comply with the planned procedures and scheduled visits of the study protocol.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Primary VL patients, admitted for treatment at the Leishmaniasis Research and Treatment Centre, Gondar University Hospital, with current standard combination therapy in eastern Africa (SSG+PM). A total of 60 VL patients is the target.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To assess the diagnostic performance of the immunological tests under evaluation for predicting cure and treatment failure at end-of-treatment assessment | At 6 month follow up
  Sensitivity, specificity, positive and negative predictive values will be reported
To assess the diagnostic performance of the molecular tests under evaluation for predicting cure and treatment failure at end-of-treatment assessment | At 6 month follow up
  Sensitivity, specificity, positive and negative predictive values will be reported

SECONDARY OUTCOMES:
To assess the diagnostic performance of the immunological tests under evaluation for predicting cure, treatment failure and relapse during follow-up | 17 days from treatment start
  After treatment completion Sensitivity, specificity, positive and negative predictive values will be reported
To assess the diagnostic performance of the molecular tests under evaluation for predicting cure, treatment failure and relapse during follow-up | 17 days from treatment start
  After treatment completion Sensitivity, specificity, positive and negative predictive values will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Leishmaniasis Research and Treatment Centre, Gondar University Hospital, Gonder, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided